CLINICAL TRIAL: NCT06838442
Title: Rehabilitation Exercise and Education of Airway Clearance Technique in Nontuberculous Mycobacterial Pulmonary Disease: A Prospective Cohort Study
Brief Title: Rehabilitation Exercise and Education of Airway Clearance Technique in NTM-PD: A Prospective Cohort Study
Acronym: NTM-Rehab
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Jun Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2501-949-303
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NTM-PD Pulmonary Rehabilitation Cohort: This cohort consists of adults diagnosed with nontuberculous mycobacterial pulmonary disease (NTM-PD) who will undergo pulmonary rehabilitation and airway clearance training as part of a prospective observational study. Participants will receive an 8-week biweekly pulmonary rehabilitation program, including oscillating positive expiratory pressure (OPEP) therapy, high-frequency chest wall oscillation (HFCWO), huffing and coughing techniques, breathing exercises, and aerobic/strength training. They will be monitored at baseline, during treatment, and at 2-month and 6-month follow-ups, undergoing pulmonary function tests (PFT), bacteriologic assessments, radiographic imaging (CT/X-ray), symptom evaluations, and quality of life assessments (EQ-5D-5L, CAT score). This study aims to assess the effectiveness of non-pharmacological interventions in improving respiratory function, reducing symptoms, and enhancing quality of life in NTM-PD patients.

SUMMARY:
* The goal of this observational study is to evaluate the effects of pulmonary rehabilitation and airway clearance education in adults with nontuberculous mycobacterial pulmonary disease (NTM-PD). The main questions it aims to answer are:

  * Does pulmonary rehabilitation and airway clearance training improve lung function, symptom relief, and quality of life in patients with NTM-PD?
  * Does this non-pharmacological intervention contribute to better sputum culture conversion rates?
* Participants will:

  * Undergo pulmonary rehabilitation and airway clearance training over an 8-week period (biweekly sessions).
  * Receive evaluations at baseline, during the intervention, and follow-up assessments at 2 months, 6 months, and final study visit.
  * Undergo tests including pulmonary function tests (PFT), symptom assessments, bacteriologic evaluations, radiographic imaging (CT/X-ray), and quality of life surveys (EQ-5D-5L, CAT score).
* This study aims to provide clinical evidence supporting the role of non-pharmacological treatments in the management of NTM-PD, potentially informing future treatment guidelines and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older at the time of enrollment.
* Diagnosis of nontuberculous mycobacterial pulmonary disease (NTM-PD) according to the 2020 American Thoracic Society (ATS) guidelines.
* Identification of clinically significant NTM species, including:

Mycobacterium avium / Mycobacterium intracellulare / Mycobacterium abscessus / Mycobacterium massiliense / Mycobacterium kansasii /

* Able to undergo pulmonary rehabilitation and airway clearance training as part of the study protocol.
* Willing to provide written informed consent to participate in the study.

Exclusion Criteria:

* Currently pregnant or actively breastfeeding.
* Unable to participate in pulmonary rehabilitation due to severe mobility impairment or neuromuscular disorders.
* History of massive hemoptysis or other medical conditions where airway clearance techniques may be contraindicated.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients (≥20 years old) diagnosed with nontuberculous mycobacterial pulmonary disease (NTM-PD) based on the 2020 American Thoracic Society (ATS) guidelines. Participants will be recruited from outpatient pulmonary clinics at Bundang Seoul National University Hospital. Eligible participants will undergo pulmonary rehabilitation and airway clearance training as part of a prospective observational study. The study focuses on assessing the effects of non-pharmacological interventions on lung function, symptom relief, and quality of life in patients with NTM-PD.
  The cohort will include patients with clinically significant NTM species such as Mycobacterium avium, Mycobacterium intracellulare, Mycobacterium abscessus, Mycobacterium massiliense, and Mycobacterium kansasii. Participants will undergo baseline assessment, structured rehabilitation sessions, and follow-up evaluations at 2 months and 6 months. The study aims to provide real-world clinical evidence sup
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2028-11-25 (Estimated); Study Completion 2028-11-25 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Function (FEV1 and FVC) from Baseline to 6 Months | Baseline, 2 months, 6 months
  Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) will be measured using pulmonary function tests (PFTs) at baseline, after 2 months, and at 6 months to assess improvements in lung function following pulmonary rehabilitation and airway clearance training.
Sputum Culture Conversion Rate | Baseline, 2 months, 6 months
  The percentage of participants achieving sputum culture conversion, defined as three consecutive negative mycobacterial cultures from respiratory samples collected at least one month apart, will be assessed.
6MWT | Baseline, 2 months, 6 months
  6 minute walk test distance in meters

SECONDARY OUTCOMES:
Change in Questionnaire-Bronchiectasis (QOL-B) from Baseline to 6 Months | Baseline, 2 months, 6 months
  Quality of life improvements will be assessed using Questionnaire-Bronchiectasis (QOL-B). The questionnaire comprised a total of 37 items, covering domains such as physical functioning (5 items), role functioning (5 items), vitality (3 items), emotional functioning (4 items), social functioning (4 items), health perception (4 items), respiratory symptoms (9 items), and treatment burden (3 items). Each domain score ranged from 0 to 100, with higher scores indicating better quality of life.
Change in EuroQoL 5-Dimension 5-Level (EQ-5D-5L) from Baseline to 6 Months | Baseline, 2 months, 6 months
  EuroQoL 5-Dimension 5-Level (EQ-5D-5L) includes quality of life assessments including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores can range from 11111 to 55555, with lower scores referring tobetter quality of life.
Severity of radiographic findings | Baseline, 2 months, 6 months
  High-resolution computed tomography (HRCT) and chest X-rays will be used to evaluate changes in lung structure, including bronchiectasis severity and cavitary lesions. Presence and size of cavities will be measured in chest CT, and artificial intelligenced-based scoring systems will be used to measure radiographic severity in chest X-rays.

OTHER OUTCOMES:
Change in Physical Function (Grip Strength, 4-Meter Walk Test, Sit-to-Stand Test) from Baseline to 6 Months | Baseline, 2 months, 6 months
  Physical function will be assessed using hand-grip strength measurements, a 4-meter walk test, and a sit-to-stand test to evaluate improvements in muscle strength and mobility.
Adverse Events Related to Pulmonary Rehabilitation and Airway Clearance Techniques | Throughout study period (up to 6 months)
  The incidence of adverse events such as fatigue, muscle pain, hemoptysis, and respiratory distress related to pulmonary rehabilitation interventions will be monitored and documented.
Change in body composition: bioimpeance analysis | Baseline, 2 months, 6 months
  Change in body composition will be assesed using the bioimpedance analysis. It provides resistance and reactance measured at different frequency currents, providing estimations of the body fat mass (kg), protein mass (kg), and skeletal muscle mass (kg). Volume of body water (L) and percentage of body fat (%) will be calculated as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
At this time, there is no plan to publicly share individual participant data (IPD) due to patient confidentiality and ethical considerations. However, de-identified, aggregated data may be made available upon reasonable request for collaborative research purposes, subject to appropriate ethical approvals and institutional review board (IRB) regulations. If data sharing becomes feasible, it will follow applicable regulations and data protection guidelines.